CLINICAL TRIAL: NCT05183828
Title: Association of HSD3B1 Genotype With Response to Preoperative Letrozole Therapy Among Postmenopausal Women With Estrogen-Receptor Positive (ER+) HER2/Neu-Negative (HER2-) Invasive Carcinomas of the Breast
Brief Title: Effect of HSD3B1 (1245C) Gene Mutation on Treatment of Stage I-III Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121659; NCI-2021-12428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IR10794 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Adenocarcinoma; Invasive Breast Carcinoma of No Special Type
MeSH Terms: conditions — Carcinoma, Ductal | interventions — Specimen Handling; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (letrozole) (Experimental): Patients receive letrozole PO QD for 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of saliva samples. If tumor resection occurs before or after day 22, letrozole administration must occur for a minimum of 14 days and a maximum of 70 days of total treatment.
  Interventions: Procedure: Biospecimen Collection; Drug: Letrozole; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This stage IV trial examines how a mutation in HSD3B1 (1245C) gene affects treatment of stage I-III breast cancer. This trial may help researchers determine if mutations in HSD3B1 decreases the efficacy of aromatase inhibitor therapy such as letrozole. Letrozole may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive letrozole orally (PO) once daily (QD) for 21 days in the absence of disease progression or unacceptable toxicity. If tumor resection occurs before or after day 22, letrozole administration must occur for a minimum of 14 days and a maximum of 70 days of total treatment. Patients also undergo collection of saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be female age >= 18 years.
* Postmenopausal as defined by at least one of the following:

  * Age >= 60 years;
  * Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; or serum estradiol and follicle stimulating hormone levels within the local laboratory's normal reference range for postmenopausal females;
  * Documented bilateral oophorectomy.
* Histologically confirmed diagnosis of carcinoma of the breast, clinical stage I-III.
* Minimum tumor diameter of 1.0 cm as assessed by palpation or imaging (e.g., ultrasound) and with enough tumor left after the initial diagnostic biopsy to provide tumor tissue during the planned tumor resection.
* Candidate for surgical resection.
* ER+ breast cancer (> 1% positive stained cells) based on the most recent tumor biopsy documented by a local laboratory or medical record.
* Ki67 >= 10%.
* HER2-negative breast cancer based on the most recent tumor biopsy and documented by a local laboratory or medical record. HER2-negative tumor is defined per American Society of Clinical Oncology and the College of American Pathologists guidelines, 2018.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Prior use of hormone contraceptives and replacement therapy is allowed (e.g., estrogen and/or progestin) if discontinued > 6 months prior to diagnosis. Vaginal preparations are allowed.
* Ability to take oral medication and be willing to adhere to the study intervention.

Exclusion Criteria:

* Pre-treatment tumor biopsy sample not likely to provide adequate tissue sections for biomarker assays.
* Inoperable or metastatic disease.
* Subjects who have received any prior therapy for breast cancer, including radiotherapy, surgery, and cytotoxic and endocrine treatments.
* The subject must not have had hormonal therapy for breast cancer treatment or for breast cancer prevention within 1 year prior to study enrollment. (Note: Synchronous breast, cancer (including bilateral breast cancer) at separate sites is permissible, provided the patient does not receive medical treatments for breast cancer or radiation therapy to the ipsilateral breast during the study intervention period.
* Subjects with plans to undergo neoadjuvant chemotherapy.
* Use of hormonal contraceptives within 6 months of diagnosis.
* Treatment with another investigational drug or other intervention within 28 days before the first administration of letrozole.
* History of allergic reactions/hypersensitivity attributed to compounds of similar chemical or biologic composition to letrozole or any ingredients.
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Ki67 | Before (baseline) and up to 9 months after surgery
  Will be assessed according to germline status.
Changes in Ki67 | Before (baseline) and up to 9 months after surgery
  Will be assessed according to somatic HSD3B1 (1245C) variant status.
Changes in estrogen receptor (ER)alpha | Before (baseline) and up to 9 months after surgery
  Will be assessed according to germline status.
Changes in estrogen receptor (ER)alpha | Before (baseline) and up to 9 months after surgery
  Will be assessed according to somatic HSD3B1 (1245C) variant status.
Changes in ER beta | Before (baseline) and up to 9 months after surgery
  Will be assessed according to germline status.
Changes in ER beta | Before (baseline) and up to 9 months after surgery
  Will be assessed according to somatic HSD3B1 (1245C) variant status.
Effect of HSD3B1 (1245C) variant on changes in Ki67 | Before (baseline) and up to 9 months after surgery
  Will evaluate whether androgen receptor (AR)+ modifies the effect of HSD3B1 (1245C) variant on changes in Ki67 before and after preoperative letrozole treatment, and whether this effects ER- and AR- gene expression signatures.
Expression of 3betaHSD1 | Up to 9 months after surgery
  Will compare expression of 3betaHSD1 according to HSD3B1 allele status.
Expression of intracellular androgen | Up to 9 months after surgery
  Will compare expression of intracellular androgen according to HSD3B1 allele status.
Expression of estrogen levels | Up to 9 months after surgery
  Will compare expression of estrogen levels according to HSD3B1 allele status.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan R. Flanagan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No